CLINICAL TRIAL: NCT06391216
Title: The Effect of Supplementation With Lactobacillus Helveticus R0052 and Bifidobacterium Longum R0175 Combination Probiotic on Mental Health Indices and Oral Microbiota Status in Healthy Volunteers Facing a Stressful Event
Brief Title: The Effect of Probiotic Supplementation on Mental Health in Healthy Volunteers
Acronym: ProBeMent
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of Lodz (Other)
Collaborators: Pomeranian Medical University Szczecin (Other); SANPROBI Sp. z o.o. Sp.k. (Unknown)
Responsible Party: Principal Investigator, Michal Karbownik, Associate Professor, Medical University of Lodz
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: ProBeMent
Record Dates: First submitted 2024-04-23; First posted 2024-04-30 (Actual); Last update posted 2024-07-12 (Actual); Status verified 2024-07

CONDITIONS: Healthy; Stress-related Problem; Depression; Anxiety
Keywords: Probiotics; Academic examination; Psychological stress; Depression; Anxiety
MeSH Terms: conditions — Depression; Anxiety Disorders; Stress, Psychological

STUDY DESIGN:
Intervention Model Description: Healthy medical students are assigned
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Probiotic (Experimental): Lactobacillus helveticus R0052 and Bifidobacterium longum R0175 combination probiotic - encapsulated
  Interventions: Dietary Supplement: Lactobacillus helveticus R0052 and Bifidobacterium longum R0175
- Placebo (Placebo Comparator): Mixture of potato starch and magnesium stearate (the excipients that are present in the tested product) - encapsulated
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Lactobacillus helveticus R0052 and Bifidobacterium longum R0175 — 8-week supplementation (56 days); 3 × 10^9 CFU/day
  Arms: Probiotic
Dietary Supplement: Placebo — 8-week supplementation (56 days)
  Arms: Placebo

SUMMARY:
Probiotics are "live microorganisms which when administered in adequate amounts confer a health benefit on the host". Accumulating evidence indicates their effect in mental health restoration. Beneficial neuropsychological and psychobiological effects are particularly well substantiated in clinical samples. However, it is not clearly documented whether probiotic supplementation reduces depressive and anxiety symptoms in healthy volunteers experiencing temporal deterioration in mental functioning while facing a stressful event. The combination of Lactobacillus helveticus R0052 and Bifidobacterium longum R0175 is particularly well studied in terms of its central nervous system action with significantly deciphered mechanism. As a result, this combination is particularly promising to study the effect of mental health improvement in healthy volunteers facing a stressful event.

The aim of this project is to assess the impact of a 8-week supplementation with probiotic combination of Lactobacillus helveticus R0052 and Bifidobacterium longum R0175 strains in the daily dose of 3 × 10^9 colony forming units on mental health measures and oral microbiota composition and metabolome in healthy young adults facing a psychologically stressful event. The aim will be achieved by comparing the probiotic combination supplement to placebo in a randomized triple-blind controlled trial settings with a participant allocation ratio of 1:1.

The summer academic examination session and the upcoming first take of the final exam in pharmacology at third year of medical studies will be a model of a stressful event. The participants will supplement their diets with probiotic/placebo for 8 weeks before the exam. After giving written informed consent, before the supplementation (relatively stress-free time period in terms of academic activities) the participants will provide background sociodemographic, anthropometric and psychometric data. At that time, participants will also give samples of saliva to assess cortisol and selected cytokines concentrations as well as salivary microbiome and metabolome. At the end of supplementation, a day before the final exam, participants will donate salivary samples and do psychometric tests for the second time to assess the same parameters as at the beginning of the study. Participants will also do a pre-exam test in pharmacology (not considered a formal academic assessment) as a comparator for the results of the formal examination held a day after.

ELIGIBILITY:
Inclusion Criteria:

* status of a third-year medical student at the Faculty of Medicine of the Medical University of Lodz
* age (18-30 years)
* high motivation and no formal obstacles to sit the first take of the final exam in pharmacology
* Body mass index of 18-25 kg/m2

Exclusion Criteria:

* chronic dental diseases (in particular periodontal diseases), neurological, psychiatric, cardiological, gastroenterological, endocrinological, immunological, inflammatory or infectious diseases or disorders
* psychiatric or neurological diagnosis - within the last 1 year
* immune disorders or possible immunodeficiency - within the last 5 years
* previous bariatric surgery - within the last 5 years
* hospitalization - within the last 3 months
* presence of central venous catheters
* use of enteral nutrition (feeding tube or nutritional fistula)
* pregnant or planning to become pregnant in the next 3 months
* breast-feeding
* occurrence of an allergic reaction - within the last 3 months
* hypersensitivity to potato starch or magnesium stearate
* chronic use of any medicinal products - within the last 3 months
* use of systemic antibacterial or antifungal drugs - within the last 1 month
* alcohol abuse (≥ 20 g or ≥ 40 g of alcohol per day for women and men, respectively) - within the last 3 months
* abuse of narcotic or psychotropic substances - within the last 3 months
* regular smoking of tobacco or other nicotine products, including e-cigarettes (> 5 cigarettes or equivalents per day - within the last 3 months)
* use of probiotic or prebiotic preparations - within the last 1 month
* a vegan diet or any unusual diet

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 100 (Actual)
Dates: Start 2024-05-06 (Actual); Primary Completion 2024-07-05 (Actual); Study Completion 2024-07-05 (Actual)

PRIMARY OUTCOMES:
Cortisol | Day 0, Day 55
  Salivary cortisol level measured with ELISA test
Depression symptoms under examination-related stress | Day 0, Day 55
  Depression symptoms measured with Depression Anxiety Stress Scale - 21 (DASS-21). Seven items, each scored 0 to 3 points, yielding a total between 0 and 21 points. The more points the more severe depression.
Anxiety symptoms under examination-related stress | Day 0, Day 55
  Anxiety symptoms measured with Depression Anxiety Stress Scale - 21 (DASS-21). Seven items, each scored 0 to 3 points, yielding a total between 0 and 21 points. The more points the more severe anxiety.
Stress symptoms under examination-related stress | Day 0, Day 55
  Stress symptoms measured with Depression Anxiety Stress Scale - 21 (DASS-21). Seven items, each scored 0 to 3 points, yielding a total between 0 and 21 points. The more points the more severe stress.
Performance under examination-related stress | Day 56
  Number of correctly-answered questions in the final examination in pharmacology in relation to subject knowledge assessed in the pre-exam test. 60 questions, each scored 0 or 1 point, yielding a total between 0 and 60 points. The more points the better performance under examination-related stress.

SECONDARY OUTCOMES:
Interleukin-1β (IL-1β) | Day 0, Day 55
  Salivary IL-1β level measured with ELISA test in relation to total protein concentration in saliva
Interleukin-8 (IL-8) | Day 0, Day 55
  Salivary IL-8 level measured with ELISA test in relation to total protein concentration in saliva
Microbiome | Day 0, Day 55
  Salivary microbiome assessed with 16S rRNA gene sequencing
Metabolome | Day 0, Day 55
  Salivary metabolome assessed with liquid chromatography-mass spectrometry
Mood | Day 0, Day 55
  Current mood measured with a pictogram-enhanced visual analog mood scale. A single item scored 0 to 10 points, yielding a total between 0 and 10 points. The more points the better mood.
Depression symptoms under examination-related stress (supportive measure) | Day 0, Day 55
  Depression symptoms measured with Patient Health Questionnaire - 9 (PHQ-9). Nine items, each scored 0 to 3 points, yielding a total between 0 and 27 points. The more points the more severe depression.
Anxiety symptoms under examination-related stress (supportive measure) | Day 0, Day 55
  Anxiety symptoms measured with General Anxiety Disorder - 7 (GAD-7). Seven items, each scored 0 to 3 points, yielding a total between 0 and 21 points. The more points the more severe anxiety.
Sleep quality under examination-related stress | Day 0, Day 55
  Sleep quality status measured with Pittsburgh Sleep Quality Index (PSQI). Seven components, each scored 0 to 3 points, yielding a total composite score of 0 to 21 points. The more points the more sleep difficulties.
Fatigue under examination-related stress | Day 0, Day 55
  Fatigue status measured with Fatigue Severity Scale (FSS). Nine items, each scored 1 to 7 points, yielding a total between 7 and 63 points. The more points the greater fatigue severity.

CONTACTS AND LOCATIONS:
Overall Officials: Michał S. Karbownik, PhD, Study Chair — Medical University of Lodz
Locations (1):
- Medical University of Lodz, Lodz, Poland

REFERENCES:
- [Background] Messaoudi M, Lalonde R, Violle N, Javelot H, Desor D, Nejdi A, Bisson JF, Rougeot C, Pichelin M, Cazaubiel M, Cazaubiel JM. Assessment of psychotropic-like properties of a probiotic formulation (Lactobacillus helveticus R0052 and Bifidobacterium longum R0175) in rats and human subjects. Br J Nutr. 2011 Mar;105(5):755-64. doi: 10.1017/S0007114510004319. Epub 2010 Oct 26. PMID 20974015
- [Background] Ait-Belgnaoui A, Colom A, Braniste V, Ramalho L, Marrot A, Cartier C, Houdeau E, Theodorou V, Tompkins T. Probiotic gut effect prevents the chronic psychological stress-induced brain activity abnormality in mice. Neurogastroenterol Motil. 2014 Apr;26(4):510-20. doi: 10.1111/nmo.12295. Epub 2013 Dec 30. PMID 24372793
- [Background] Ait-Belgnaoui A, Payard I, Rolland C, Harkat C, Braniste V, Theodorou V, Tompkins TA. Bifidobacterium longum and Lactobacillus helveticus Synergistically Suppress Stress-related Visceral Hypersensitivity Through Hypothalamic-Pituitary-Adrenal Axis Modulation. J Neurogastroenterol Motil. 2018 Jan 30;24(1):138-146. doi: 10.5056/jnm16167. PMID 29291614
- [Background] Chao L, Liu C, Sutthawongwadee S, Li Y, Lv W, Chen W, Yu L, Zhou J, Guo A, Li Z, Guo S. Effects of Probiotics on Depressive or Anxiety Variables in Healthy Participants Under Stress Conditions or With a Depressive or Anxiety Diagnosis: A Meta-Analysis of Randomized Controlled Trials. Front Neurol. 2020 May 22;11:421. doi: 10.3389/fneur.2020.00421. eCollection 2020. PMID 32528399
- [Background] Karbownik MS, Kreczynska J, Kwarta P, Cybula M, Wiktorowska-Owczarek A, Kowalczyk E, Pietras T, Szemraj J. Effect of Supplementation with Saccharomyces Boulardii on Academic Examination Performance and Related Stress in Healthy Medical Students: A Randomized, Double-Blind, Placebo-Controlled Trial. Nutrients. 2020 May 19;12(5):1469. doi: 10.3390/nu12051469. PMID 32438624